CLINICAL TRIAL: NCT00704431
Title: An Open Label, Single Session Study to Collect Tolerability Information Following Repeat Dosing of Darapladib in Healthy Adult Subjects
Brief Title: A Study With Darapladib to Collect Tolerability Information
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPL111814
Record Dates: First submitted 2008-06-20; First posted 2008-06-24 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Atherosclerosis
Keywords: SB-480848; darapladib; tolerability
MeSH Terms: conditions — Atherosclerosis | interventions — darapladib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- darapladib (Experimental): darapladib
  Interventions: Drug: SB-480848 (darapladib)

INTERVENTIONS:
Drug: SB-480848 (darapladib) — 160 mg darapladib

SUMMARY:
Subjects will receive their first dose of darapladib in the clinical research unit (CRU), and the remaining 9 days of dosing will occur at home. Subjects will record any adverse events throughout the dosing period in a paper diary. Subjects will return to the CRU 10-14 days after the last dose of darapladib for a follow-up visit. The total study duration for each subject including the screening, treatment and follow-up periods will be approximately 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and ECG.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of:

  * Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea
  * Child-bearing potential and agrees to use one of the contraception methods listed in the protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow-up visit.
* Body weight >= 50 kg and BMI within the range 19 - 30 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* History of drug abuse.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* History of anaphylaxis, anaphylactoid reactions and severe allergic responses.
* History of adult asthma manifested by bronchospasms in the past 6 months or currently taking regular anti-asthmatic medication.
* Currently receiving oral or injectable strong CYP3A4 inhibitor(s).
* Consumption of grapefruit or grapefruit juice within 7 days prior to first dose of study medication.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum hCG test at screening.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Adverse events as reported by subjects. | From dosing through to follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, King of Prussia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: LPL111814 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: LPL111814 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: LPL111814 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: LPL111814 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: LPL111814 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: LPL111814 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register